CLINICAL TRIAL: NCT02831790
Title: The Fontan Education Study: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: The Fontan Education Study
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-05

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention (Experimental): Participants in the intervention group will have access to the 3 teaching videos, ~3:30-5:00 minutes in duration each, beginning several weeks prior to the preadmission clinic (as soon as written consent is obtained).
  Interventions: Other: Fontan Education Videos
- Usual Care (No Intervention): Participants in the usual care will not be offered an intervention and will not be made aware of the existence of the teaching videos.

INTERVENTIONS:
Other: Fontan Education Videos — The intervention will consist of three brief (~5 minute) professionally-developed whiteboard videos, available online. The videos will feature lay language at a grade 7 level or below and will be engaging. Topics are based on key findings of the Family Resilience Study, namely:
  1. Stress reactions in children and parents post Fontan. This video will be supplemented with existing resources on the topic.
  2. Anticoagulation
  3. Prolonged pleural drainage
  Arms: Educational Intervention

SUMMARY:
The Fontan Education Study is a cluster randomized controlled trial evaluating the impact of a novel education program in combination with usual care, versus usual care alone, on preparing parents of children undergoing Fontan surgery for the challenges of the postoperative course.

ELIGIBILITY:
Inclusion Criteria:

* children who are planned to undergo Fontan surgery within 4-6 weeks and their parent(s)/guardian(s)

Exclusion Criteria:

* parents with < grade 6 level of English reading.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Parent's State Anxiety Inventory (STAI)-State score preoperatively | within 1 week preceding surgery
  The primary endpoint is the parent's STAI-State score within 1 week preceding surgery.

SECONDARY OUTCOMES:
STAI-State score postoperatively | 1 week and 1 month postoperatively
  Parent STAI-State score 1- week and 1-month postoperatively
Post-Hospital Behaviour Questionnaire (PHBQ) score postoperatively | 1 week and 1 month postoperatively
  child's PHBQ score 1 week and 1 month postoperatively

OTHER OUTCOMES:
Semi-structured interviews postoperatively | 1 Month Postoperatively
  Semi-structured interviews will be conducted by a trained qualitative interviewer who works with a team member and has extensive experience with parents.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Mackie, MD, SM, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada